CLINICAL TRIAL: NCT04797143
Title: Impact of a Multidisciplinary Consultation Program on Drug Adherence in First Oral Anticancer Treatment
Acronym: IMPAM
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0023
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Multidisciplinary Consultation Program; Adherence to Oral Anticancer Treatment; Drug Related Toxicity; Securing Medication Management
Keywords: Multidisciplinary consultation program; adherence to oral anticancer treatment; drug related toxicity; securing medication management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: patients in control group receive standard care
- intervention group: intervention group after implementation of a MCP
  Interventions: Device: multidisciplinary consultation program

INTERVENTIONS:
Device: multidisciplinary consultation program — The multidisciplinary consultation program (MCP) was divided into 3 steps: the first step involved a consultation with an oncologist, the second step involved a consultation with an oncology pharmacist, and the third step involved a meeting with a coordinating nurse (CN). The CN put in place a regular telephone follow-up with the patient, a few days later (7 to 15 days), to ensure adherence and tolerance of the oral anticancer treatment (OAT).
  Groups: intervention group

SUMMARY:
Oncology management has changed dramatically over the last decade with the approval and rapid adoption of newly targeted oral oncology medications. The movement to oral oncology medications has altered the balance of risks and adverse effects (AEs) in the treatment of cancer care. These treatments are associated with a different constellation of AEs and drug interactions. Patients receiving treatment with oral anticancer treatment (OAT) encounter several barriers to adherence, which may include limited access to specialty medications, severe adverse effects, complex medication regimens, and special handling precautions. Medication nonadherence not only reduces the efficacy of drug therapy but also has the potential to increase healthcare expenditures due to disease-related hospitalizations. The purpose of this study is to evaluate the drug adherence in cancer patients, using the medication possession ratio (MPR), before and after the implementation of a multidisciplinary consultation program (MCP), on initiation of OAT.

ELIGIBILITY:
Inclusion Criteria:

* French speaking patients with a newly diagnosed or relapsed cancer, regardless of location and introduction of oral anticancer treatment

Exclusion Criteria:

* patients treated with hormone therapy only
* Patient with severe psychiatric disorders
* patient who does not speak the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with standard treatment or after implementation of a MCP The MCP was divided into 3 steps: the first step involved a consultation with an oncologist, the second step involved a consultation with an oncology pharmacist, and the third step involved a meeting with a coordinating nurse CN. The CN put in place a regular telephone follow-up with the patient, a few days later (7 to 15 days), to ensure adherence and tolerance of the OAT.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
medication possession ratio (MPR) | two months
  The MPR makes it possible to determine the percentage of days of treatment covered by pharmacy dispensing. A patient is generally considered observant if MPR is greater than or equal to 80%.
medication possession ratio (MPR) | one year
  The MPR makes it possible to determine the percentage of days of treatment covered by pharmacy dispensing. A patient is generally considered observant if MPR is greater than or equal to 80%.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No